CLINICAL TRIAL: NCT02693223
Title: Get With the Guidelines-Stroke Registry
Acronym: GWTG-Stroke
Status: Recruiting | Type: Observational
Sponsor: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: GWTG Stroke program — Evidence based recommended therapies and counseling prior to hospital discharge.

SUMMARY:
Get With The Guidelines-Stroke is a program for improving the quality of care for patients hospitalized with stroke by promoting consistent adherence to the latest evidence-based clinical practice guidelines.

DETAILED DESCRIPTION:
Get With The Guidelines®-Stroke is an in-hospital program for improving stroke care by promoting consistent adherence to the latest scientific treatment guidelines. Since its initiation in 2003, 2,637 hospitals have entered 3,892,063 patient records into the Get With The Guidelines-Stroke database. Numerous published studies demonstrate the program's success in achieving measurable patient outcome improvements.

Achievement measures tracked through the Get With The Guidelines®-Stroke:

* IV rT-PA arrive by 3.5 hour, treat by 4.5hour
* Early antithrombotics
* VTE prophylaxis
* Antithrombotics at or by discharge
* Anticoagulation for Afib/Aflutter at or by discharge
* Smoking cessation at or by discharge
* Intensive Statin Therapy

Quality measures tracked through the Get With The Guidelines®-Stroke:

* Dysphagia screen
* Time to intravenous thrombolytic therapy-60 min
* NIHSS reported
* Stroke education at or by discharge
* Rehabilitation considered at or by discharge
* LDL Documented

Additional measures collected by Get With The Guidelines®-Stroke can be viewed at: https://www.heart.org/en/professional/quality-improvement/get-with-the-guidelines/get-with-the-guidelines-stroke/get-with-the-guidelines-stroke-patient-management-tool

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with a diagnosis of Ischemic stroke or transient ischemic attack, Subarachnoid hemorrhage, Intracerebral hemorrhage, or Stroke not otherwise specified to the hosptials.

Exclusion Criteria:

* Patients who do not have a diagnosis of Ischemic stroke or transient ischemic attack, Subarachnoid hemorrhage, Intracerebral hemorrhage, or Stroke not otherwise specified.
* Patients under age of 18

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Ischemic stroke or transient ischemic attack, Subarachnoid hemorrhage, Intracerebral hemorrhage, or Stroke not otherwise specified.
Sampling Method: Probability Sample
Enrollment: 3892063 (Estimated)
Dates: Start 2003-01; Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 6 days - mean for length of hospitalization for Stroke patients
Modified Rankin Scale at Discharge | 6 days - mean for length of hospitalization for Stroke patients
  Patients grouped by Modified Rankin Scale at discharge
Risk-Adjusted Mortality Ratio (for Ischemic-Only and Ischemic and Hemorrhagic models) | 30 days post discharge from hospital
  A ratio comparing the actual in-hospital mortality rate to the risk-adjusted expected mortality rate.

CONTACTS AND LOCATIONS:
Overall Officials: Javed Butler, MD, Study Director — American Heart Association
Locations (1):
- Amy Bennett, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mulder MJ, van Oostenbrugge RJ, Dippel DW; MR CLEAN Investigators. Letter by Mulder et al Regarding Article, "2015 AHA/ASA Focused Update of the 2013 Guidelines for the Early Management of Patients With Acute Ischemic Stroke Regarding Endovascular Treatment: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association". Stroke. 2015 Nov;46(11):e235. doi: 10.1161/STROKEAHA.115.010913. Epub 2015 Oct 8. No abstract available. PMID 26451021
- [Result] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637
- [Result] Meschia JF, Bushnell C, Boden-Albala B, Braun LT, Bravata DM, Chaturvedi S, Creager MA, Eckel RH, Elkind MS, Fornage M, Goldstein LB, Greenberg SM, Horvath SE, Iadecola C, Jauch EC, Moore WS, Wilson JA; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Functional Genomics and Translational Biology; Council on Hypertension. Guidelines for the primary prevention of stroke: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Dec;45(12):3754-832. doi: 10.1161/STR.0000000000000046. Epub 2014 Oct 28. PMID 25355838
- [Result] Saver JL, Carroll JD, Smalling R, Thaler D. Letter by Saver et al regarding article, "Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association". Stroke. 2015 Apr;46(4):e85-6. doi: 10.1161/STROKEAHA.115.007311. Epub 2015 Mar 5. No abstract available. PMID 25744518
- [Result] Powers WJ, Derdeyn CP, Biller J, Coffey CS, Hoh BL, Jauch EC, Johnston KC, Johnston SC, Khalessi AA, Kidwell CS, Meschia JF, Ovbiagele B, Yavagal DR; American Heart Association Stroke Council. 2015 American Heart Association/American Stroke Association Focused Update of the 2013 Guidelines for the Early Management of Patients With Acute Ischemic Stroke Regarding Endovascular Treatment: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Oct;46(10):3020-35. doi: 10.1161/STR.0000000000000074. Epub 2015 Jun 29. PMID 26123479